CLINICAL TRIAL: NCT07350512
Title: Investigating the Effect of Glucagon on Cognitive Function and Cerebral Glucose Metabolism in Humans: A Pilot Study
Brief Title: Investigating the Acute Effects of Increasing Alanine Exposure in Healthy Participants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nicolai Jacob Wewer Albrechtsen (Other)
Responsible Party: Sponsor-Investigator, Nicolai Jacob Wewer Albrechtsen, Principal Investigator, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GluCoMet_stepwise alanine
Record Dates: First submitted 2026-01-09; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Glucose Metabolism; Glucagon
Keywords: Alanine; glucagon; glucose metabolism
MeSH Terms: interventions — Alanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Alanine infusion (Experimental)
  Interventions: Other: alanine

INTERVENTIONS:
Other: alanine — A three-hour intravenous infusion with alanine with increasing infusion rate (from 1.4 μmol/kg/min and to 28 μmol/kg/min)

SUMMARY:
In this study the investigators will investigate the acute effects of increasing alanine exposure on metabolic parameters in healthy participants.

Participants will participate in one study day. After initial baseline blood samples, a three-hour intravenous infusion with glucagon will be initiated. The infusion rate will be increased every 30 minutes.

DETAILED DESCRIPTION:
Two peripheral catheters will be placed in the antecubital vein of each arm for infusion of L-alanine and blood sampling respectively. The infusion rate of alanine will start at 1.4 μmol/kg/min and increase every 30 minutes over a 3-hour period, up to a maximum of 28 μmol/kg/min. The study day will last approximately 4 hours, and a maximal blood volume of 130 ml will be collected. Blood samples for the analysis of plasma glucagon, glucose, insulin, C-peptide etc. will be drawn every 15 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding the participant information and signing the consent form
* Between 25 and 70 years of age at the time of screening
* Body mass index (BMI) ≤ 25 kg/m2 at the time of screening

Exclusion Criteria:

* Enrolment in other research projects that might interfere with the study
* Diabetes diagnosis (type 1 and 2)
* Pregnancy or breastfeeding
* Use of medications which, in the opinion of the investigator, may jeopardise participant's safety or compliance with the protocol
* Impaired liver function defined as either alanine aminotransferase (ALAT) and/or aspartate aminotransferase (ASAT) ≥ 2 times normal values
* Kidney disease defined as serum creatinine levels ≥ 126 μmol/L for male and ≥ 111 μmol/L for female
* Inadequately treated blood pressure at screening defined as repeated resting blood pressure outside the range 90-150 mmHg for systolic and 50-100 mmHg for diastolic
* Active or recent malignant disease
* Current or history of severe alcohol use or drug/chemical abuse as per investigator's judgement
* Any chronic disorders or severe diseases which, in the opinion of the investigator, might jeopardise participant's safety or compliance with the protocol

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-01-20 (Estimated)

PRIMARY OUTCOMES:
Threshold alanine infusion rate for stimulation of plasma glucagon | Baseline and every 30 minutes during the 0-180 min infusion period.
  Lowest alanine infusion rate (µmol/kg/min) at which plasma glucagon concentration is significantly higher than baseline during a 3-hour stepwise alanine infusion (six 30-minute steps from 1.4 to 28 µmol/kg/min).

SECONDARY OUTCOMES:
Change in plasma glucose during stepwise alanine infusion | Baseline and every 30 minutes during the 0-180 min infusion period.
  Plasma glucose concentration (mmol/L) measured at baseline and every 30 minutes during a 3-hour stepwise alanine infusion (1.4-28 µmol/kg/min), analyzed as absolute values and change from baseline.
Change in plasma follicle-stimulating hormone (FSH) during stepwise alanine infusion | Baseline and every 30 minutes during the 0-180 min infusion period.
  Plasma follicle-stimulating hormone (FSH) concentration (IU/L) measured at baseline and at the end of the 3-hour stepwise alanine infusion to explore acute effects on pituitary gonadotropin secretion.
Change in plasma luteinizing hormone (LH) during stepwise alanine infusion | Baseline and every 30 minutes during the 0-180 min infusion period.
  Plasma luteinizing hormone (LH) concentration (IU/L) measured at baseline and at the end of the 3-hour stepwise alanine infusion to explore acute effects on pituitary gonadotropin secretion.
Change in plasma cortisol during stepwise alanine infusion | Baseline and every 30 minutes during the 0-180 min infusion period.
  Plasma cortisol concentration (nmol/L) measured at baseline and every 60 minutes during the 3-hour stepwise alanine infusion to assess activation of the hypothalamic-pituitary-adrenal axis.
Change in plasma triglycerides during stepwise alanine infusion | Baseline and every 30 minutes during the 0-180 min infusion period.
  Plasma triglyceride concentration (mmol/L) measured at baseline and at the end of the 3-hour stepwise alanine infusion to evaluate acute effects on lipid metabolism.
Change in plasma urea during stepwise alanine infusion | Baseline and every 30 minutes during the 0-180 min infusion period.
  Plasma urea (carbamide) concentration (mmol/L) measured at baseline and at the end of the 3-hour stepwise alanine infusion to assess short-term effects on nitrogen metabolism.
Change in plasma alanine aminotransferase (ALAT) during stepwise alanine infusion | Baseline and every 30 minutes during the 0-180 min infusion period.
  Plasma alanine aminotransferase (ALAT/ALT) activity (U/L) measured at baseline and at the end of the 3-hour stepwise alanine infusion to assess acute changes in liver enzyme levels.
Change in plasma C-peptide during stepwise alanine infusion | Baseline and every 30 minutes during the 0-180 min infusion period.
  Plasma C-peptide concentration (pmol/L) measured at baseline and every 30 minutes during a 3-hour stepwise alanine infusion, analyzed as absolute values and change from baseline.
Change in plasma insulin during stepwise alanine infusion | Baseline and every 30 minutes during the 0-180 min infusion period.
  Plasma insulin concentration (pmol/L) measured at baseline and every 30 minutes during a 3-hour stepwise alanine infusion, analyzed as absolute values and change from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai Jacob Wewer Albrechtsen, MD PhD, Principal Investigator — Department of Clinical Biochemistry, Copenhagen University Hospital - Bispebjerg and Frederiksberg Hospital, Copenhagen, Denmark
Locations (1):
- Department of Clinical Biochemistry, Copenhagen University Hospital - Bispebjerg and Frederiksberg, Copenhagen, Denmark